CLINICAL TRIAL: NCT03496857
Title: Effect of LED Photobiomodulation on Analgesia During Labor: a Randomized Clinical Trial
Brief Title: Effect of LED Photobiomodulation on Analgesia During Labor
Acronym: EPAL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Lara Jansiski Motta, Principal Investigator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PhotobioLabor01
Record Dates: First submitted 2018-03-28; First posted 2018-04-12 (Actual); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Labor Pain
Keywords: labor pain
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Intervention Model Description: RANDOMIZED CLINICAL TRIAL
Who Masked: Outcomes Assessor
Masking Description: Statistic evaluation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Photobiomodulation analgesia (Experimental): LED therapy sessions will be held in the pre-labor room. The patient who will undergo analgesia and the professional responsible for placing the LED plate on the patient's back, between T10 and L2, will be present at the time of the intervention. The LED plate will be covered with clear disposable plastic (PVC) to avoid cross-contamination and ensure hygiene. During the interventions, the patient will be allowed to choose the position that is the most comfortable for her.
  Three 10-min LED applications will be performed when the patient has a cervical dilatation of 4-5, 6-7, and 8-9 cm. Data on the level of pain, characteristics of the membrane (intact or damaged), heart rate, cardiotocography, and uterine dynamics will be collected after each intervention.
  Interventions: Device: Light emitting diode
- bath therapy (Active Comparator): The method of analgesia with the bath therapy will be performed using a hot shower at 37°C for 10 min. After showering the entire body or the back for 5 min, the participants will be allowed to direct the water flow to any area of the body that feels the most comfortable and to adjust the temperature themselves for improved comfort. Bath therapy will be performed at three time points during labor: at cervical dilatation of 4-5 cm, 6-7 cm, and 8-9 cm. Data on the level of pain, membrane characteristics (intact or damaged), heart rate, cardiotocography, and uterine dynamics will be collected after the bath therapy by performing the same measurements used in the intervention group.
  Interventions: Other: Bath Therapy

INTERVENTIONS:
Device: Light emitting diode — Three 10-min LED applications will be performed when the patient has a cervical dilatation of 4-5, 6-7, and 8-9 cm. Data on the level of pain, characteristics of the membrane (intact or damaged), heart rate, cardiotocography, and uterine dynamics will be collected after each intervention.
  Arms: Photobiomodulation analgesia
Other: Bath Therapy — The method of analgesia with the bath therapy will be performed using a hot shower at 37°C for 10 min. After showering the entire body or the back for 5 min, the participants will be allowed to direct the water flow to any area of the body that feels the most comfortable and to adjust the temperature themselves for improved comfort. Bath therapy will be performed at three time points during labor: at cervical dilatation of 4-5 cm, 6-7 cm, and 8-9 cm. Data on the level of pain, membrane characteristics (intact or damaged), heart rate, cardiotocography, and uterine dynamics will be collected after the bath therapy by performing the same measurements used in the intervention group.
  Arms: bath therapy

SUMMARY:
The aim of this study is to valuate the effects of LED photobiomodulation on analgesia during labor.ight-emitting diode (LED) photobiomodulation is an effective and noninvasive alternative to pharmacological methods.n total, 60 women in labor admitted to a public maternity hospital will be selected for a randomized controlled trial. The participants will be randomized into two groups: intervention group [analgesia with LED therapy (n = 30)] and control group [analgesia with bath therapy (n = 30)].

DETAILED DESCRIPTION:
Background: Labor pain is one of the most intense pains experienced by women, which leads to an increase in the number of women opting to undergo a cesarean delivery. Pharmacological and nonpharmacological analgesia methods are used to control labor pain. Epidural analgesia is the most commonly used pharmacological analgesia method. However, it may have side effects on the fetus and the mother. Light-emitting diode (LED) photobiomodulation is an effective and noninvasive alternative to pharmacological methods.

Objectives: To evaluate the effects of LED photobiomodulation on analgesia during labor.

Methods: In total, 60 women in labor admitted to a public maternity hospital will be selected for a randomized controlled trial. The participants will be randomized into two groups: intervention group [analgesia with LED therapy (n = 30)] and control group [analgesia with bath therapy (n = 30)]. The perception of pain will be assessed using the visual analogue scale (VAS), with a score from 0 to 10 at baseline, i.e., before the intervention. In both the groups, the procedures will last 10 min and will be performed at three time points during labor: during cervical dilation of (1) 4-5 cm, (2) 6-7 cm, and (3) 8-9 cm. At all three time points, pain perception will be evaluated using VAS shortly after the intervention. In addition, the evaluation of membrane characteristics (intact or damaged), heart rate, uterine dynamics, and cardiotocography will be performed at all time points.

Expected outcomes: The use of LED photobiomodulation will have an analgesic effect superior to that of the bath therapy.

ELIGIBILITY:
Inclusion Criteria:

* women who request analgesia during labor
* nulliparous and multiparous
* women with term gestation
* women without previous diseases, including diabetes, neurological diseases.

Exclusion Criteria:T

* women whose labor is induced with medications;
* women who request drug analgesia during labor;
* women who undergo cesarean delivery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-03-28 (Actual); Primary Completion 2018-08-31 (Estimated); Study Completion 2018-11-20 (Estimated)

PRIMARY OUTCOMES:
Labor pain | 20 minutes
  Visual Analogue Scale Pain

CONTACTS AND LOCATIONS:
Overall Officials: Lara Motta, PhD, Principal Investigator — Nove de Julho University
Locations (1):
- Lara Motta, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Traverzim MA, Sobral APT, Fernandes KPS, de Fatima Teixeira Silva D, Pavani C, Mesquita-Ferrari RA, Horliana ACRT, Gomes AO, Bussadori SK, Motta LJ. The Effect of Photobiomodulation on Analgesia During Childbirth: A Controlled and Randomized Clinical Trial. Photobiomodul Photomed Laser Surg. 2021 Apr;39(4):265-271. doi: 10.1089/photob.2020.4976. Epub 2021 Mar 23. PMID 33760671